CLINICAL TRIAL: NCT01257152
Title: Screening MRI for Cancer Recurrence in Patients Treated With Breast Conserving Therapy
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: Screening MR for Recurred BrCa
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Breast Neoplasms; Neoplasm Recurrence, Local
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, multicenter study:

* Primary objective: to assess the diagnostic yield of screening MRI compared to physical examination, mammography or ultrasonography in the detection of recurrence in patients treated with breast conserving therapy
* Secondary objective: to describe the size, type, grade, and nodal status of cancers seen only on MRI and to estimate the rate of benign biopsies and short interval follow-up induced only by MRI in this population.

DETAILED DESCRIPTION:
* Patients treated with breast conserving therapy will be followed for recurrence in the ipsilateral or contralateral breast by physical examination every six month and imaging studies performed annually.
* The imaging including mammography, physician-performed bilateral whole breast ultrasonography and a dynamic breast MRI with gadolinium-containing contrast medium will be performed according to a standard protocol. Interpretation will be conducted independently and classified according to the Breast Imaging Reporting and Data System (BI-RADS) by experienced radiologists.
* Definitive information about the presence of malignancy will be obtained by biopsy directed by the imaging method best depicting the lesion with 14-g or 11-g needle devices or needle localized excision. The absence of breast cancer was determined by means of biopsy, the absence of positive findings on repeat imaging and clinical examination, or both at follow-up.
* After three rounds of annual screening, the diagnostic yield of screening MRI compared to physical examination, mammography or ultrasonography will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 20 years in age;
* Women who underwent breast-conserving surgery for invasive breast cancer, whose final margins were negative and who finished radiation therapy at least 6 months prior to this study;
* No history of breast biopsy of the breast within 6 months prior to this study;
* Signed study-specific informed consent prior to registration;
* Has not had contralateral mastectomy;
* No known metastatic disease;
* Not pregnant or lactating;
* No present signs or symptoms of breast cancer [no palpable mass(es), bloody or spontaneous clear nipple discharge, axillary mass, or abnormal skin changes in the breast(s) or nipple(s)].
* No contraindications to MRI examination.
* No prior MRI, US or mammography within the 6 months prior to the study.

Exclusion Criteria:

* Had a screening contrast-enhanced breast MRI within the past 24 months or diagnostic contrast-enhanced MRI on any study breasts within the past 12 months;
* Had breast surgery and/or a core biopsy on the study breast(s) performed within the prior 6 months on the study
* Currently receiving chemotherapy [with exception to participant with personal history of cancer, and on chemoprevention with Tamoxifen, Evista (Raloxifene), Arimidex (Anastrozole), Aromasin (Exemestane) or other aromatase inhibitor];
* Participant with severely impaired renal function with estimated glomerular filtration rate (GFR) < 30 mL/min/1.73m2 and/or on dialysis.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Breast cancer patients undergoing conservation surgery and radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2010-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of screening breast MRI | Three years after the first screening MRI

SECONDARY OUTCOMES:
Sensitivity, specificity, negative predictive value, and positive predictive value of screening mammography, ultrasonography, and MRI | Three years after the first screening examinations

OTHER OUTCOMES:
Complications of the MRI contrast agents | Three years after the first screening MRI

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, M.D., Ph.D., Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea